CLINICAL TRIAL: NCT00804479
Title: Unblinded, Multicenter, Prospective Follow-up of Long-term Consequences of Initiating Patients With Parkinson's Disease on Either Pramipexole or Levodopa.
Brief Title: The Long Term Impact of Initiating Pramipexole Versus Levodopa in Early Parkinson's Disease (CALM-PD Cohort Study)
Acronym: CALM-PD Cohort
Status: Terminated | Type: Observational
Why Stopped: Funding for the CALM-PD Cohort Study was terminated by sponsor.
Sponsor: University of Rochester (Other)
Collaborators: Pharmacia Corp. (Peapack, NJ) (Unknown); Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Robert Holloway, Professor, University of Rochester
Other Study IDs: PPXAPD-0072-138; RSRB #09283
Record Dates: First submitted 2008-12-04; First posted 2008-12-08 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment: Available 301 subjects enrolled in CALM-PD Available 82 subjects enrolled in CALM-PD imaging substudy
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention.

SUMMARY:
To determine the long-term consequences (8 years) of initiating patients with Parkinson's disease on either pramipexole or levodopa. We hypothesize that patients initiating therapy with pramipexole compared with levodopa will demonstrate less self-reported disability as measured by the Modified Schwab and England (S/E) scale 8 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Available 301 subjects enrolled in the CALM-PD study.

Exclusion Criteria:

* Those not enrolled in the CALM-PD study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Available 301 subjects enrolled in CALM-PD
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2002-01; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
We hypothesize that patients initiating therapy with pramipexole compared with levodopa will demonstrate less self-reported disability as measured by the Modified Schwab and England. | 8 years from date randomized in CALM study

SECONDARY OUTCOMES:
Our secondary specific aim is to develop and estimate a structural model that will allow us to uncover the causal pathways through which treatments effect outcomes. | 8 years from randomization of CALM-PD study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Parkinson Study Group CALM Cohort Investigators. Long-term effect of initiating pramipexole vs levodopa in early Parkinson disease. Arch Neurol. 2009 May;66(5):563-70. doi: 10.1001/archneur.66.1.nct90001. PMID 19433655